CLINICAL TRIAL: NCT06414200
Title: Nutritional Care After Hospital Discharge
Brief Title: Nutritional Care After Discharge in Children Term Born-18years Old
Acronym: NutriCAD
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Erasmus Medical Center (Other)
Responsible Party: Principal Investigator, S.C.A.T Verbruggen, Principal Investigator, Erasmus Medical Center
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: NL84484.078.23
Record Dates: First submitted 2024-05-02; First posted 2024-05-16 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Malnutrition, Child
Keywords: Nutritional care; After discharge; Pediatric
MeSH Terms: conditions — Child Nutrition Disorders

STUDY DESIGN:
Intervention Model Description: Multicentre study. It will be executed in an academic and five non-academic hospitals throughout The Netherlands. Due to the nature of the intervention, which involves changes to the provision of care and interaction between participants, there is a risk of cross-contamination within centers. Therefore, to avoid contamination of current practice, the stepped wedge cluster randomized controlled trial design was selected. This implies that all participating centers ('clusters') start with standard care (usual care). Subsequently, randomization will determine in which order the centers will begin with the NutriCAD intervention. In the end, all centers will have crossed over to be exposed to the NutriCAD intervention
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group/usual care group (No Intervention): The usual care as given at that moment in that hospital. The group to compare the intervention with.
- Intervention group (Active Comparator): The intervention consists of a tailored nutritional follow-up plan, including a parent empowerment program, made by a multidisciplinary support team (primarily responsible clinician, dietician, psychologist and, if indicated, a speech therapist). At discharge and follow-up at 6, 12 and 18 weeks after discharge, food diaries (including growth) and questionnaires* relating to feeding behaviour and parental stress are filled out by parents/caregivers.
  Interventions: Other: multidisciplinary structured tailored made nutritional advice

INTERVENTIONS:
Other: multidisciplinary structured tailored made nutritional advice — The goal is a structured follow-up after discharge. Parents need to fill in questionnaires about eating behavior en feeding difficulties about their child. They also need to fill in a questionnaire about their stress. Together with their nutritional intake (3-days food diary) and growth a tailor-made nutritional plan is made. All the information I showed in a dashboard and discussed it with their dietitian. Who discusses this information in a multi-disciplinary team (pediatrician, psychologist and if needed a speech therapist).
  Arms: Intervention group

SUMMARY:
The goal of this stepped wedge cluster randomized trial is to compare nutritional care after discharge to an intervention in children term born - 18 years old discharged with newly initiated nutritional care.

The main question it aims to answer is:

To investigate whether a tailored nutritional care follow-up program in children who are being discharged from the hospital with nutritional support improves nutritional intake and status as well as feeding behavior and quality of life (QoL) in children and their parents. Furthermore, the effect on parental stress, anxiety, depression, and post-traumatic stress (PTSD) as well as QoL will be assessed with and without a tailored nutritional care follow-up program

DETAILED DESCRIPTION:
All subjects, both in the usual care and intervention group, will be treated with the standard nutritional protocols of these individual hospitals during hospitalization. After hospital discharge, the treatments of the intervention and the control group will entail the procedures as described below.

Intervention group The intervention consists of a tailored nutritional follow-up plan, including a parent empowerment program, made by a multidisciplinary support team (primarily responsible clinician, dietician, psychologist and, if indicated, a speech therapist). At discharge and follow-up at 6, 12 and 18 weeks after discharge, food diaries (including growth) and questionnaires* relating to feeding behaviour and parental stress are filled out by parents/caregivers.

One week before the planned outpatient visit of the patient and their parents, questionnaires will be sent with preferred software available in ErasmusMC ICT infrastructure through e-mail. The findings gathered from these nutritional data and questionnaires will be visualized on a dashboard (visible to parents and the caregivers) to discuss and help resolve the most relevant problems with the parents during the follow-up moments. During the outpatient visit, the growth and body composition of the child will also be assessed.

The nutritional support team will discuss the outcomes of the questionnaires and make tailored advice based on the problems parents have reported. The dietician will discuss this tailored advice with the children and/or parents based on the growth, the nutritional intake of the child, and the problems parents have reported regarding the feeding behaviour of the child and their parental distress. Subsequently, the dietician will provide recommendations and psychoeducation to parents and/or patients in order to improve the nutritional status.

At 6 months after discharge follow/up measurements such as, growth, duration and frequency of nutritional support, food diary, feeding behaviour of the child, QoL of the child, parental stress and QoL will be gathered.

Evaluation and treatment other than follow-up at 6, 8 and 12 weeks after discharge with one of the health care professionals are on indication and data will not be collected.

The intervention differs from the usual care, because follow-up is at standard time periods. In the usual care this is not regulated. Nutritional support is given in a multidisciplinary team including a psychologist, but in the pilot study we saw collaboration with the pediatrician and speech therapist only. In the intervention we also focuses on parenteral stress, which is new and different from usual care.

Usual care group Nutritional advice in the usual care group will be given after discharge and follow-up according to standard practices. At 6 months after discharge an evaluation will be done equal to the intervention group. To collect information about the number of readmissions to the hospital and reason of admission, visits to a health-care provider, and growth parameters parents are asked to fill in a logbook to collect this data between discharge and 6 months follow-up. This method has been chosen because these are parameters that are difficult to remember at the visit 6 months after discharge.

*The following age-adjusted and validated questionnaires will be used to assess emotional functioning, the pediatric feeding disorders, and parenteral stress:

ELIGIBILITY:
Inclusion Criteria:

* Children term born neonates till 18 years old
* Admitted with newly initiated nutritional support(oral and/or enteral nutritional support) during hospitalization
* Nutritional Support continues at home after discharge.

Exclusion Criteria:

* Children with existing nutritional support upon admission
* Children in need of parenteral nutrition at discharge
* Children with DSM-5 diagnosed feeding disorders such as anorexia
* Absence of written informed consent

Ages: 7 Days to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 260 (Estimated)
Dates: Start 2024-12-01 (Estimated); Primary Completion 2026-03-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Weigth | From enrollment until 6 months after discharge
  in kilograms and z-scores
Height | From enrollment until 6 months after discharge
  in meters and z-scores
Head circumference | From enrollment until 6 months after discharge
  in centimeters and z-scores
Mid-upper arm circumference | From enrollment until 6 months after discharge
  in centimeters and z-scores
Length in children <2 years of age | From enrollment until 6 months after discharge
  in centimeters and z-scores

SECONDARY OUTCOMES:
Body composition | From enrollment until 6 months after discharge
  Fat mass, Fat free mass
Duration and frequency of nutritional support | From enrollment until 6 months after discharge
  Time (weeks), frequency per day
Dependency on nasogastric tube feeding | From enrollment until 6 months after discharge
  Yes/No and intermitted or portions
Nutritional requirements and intake | From enrollment until 6 months after discharge
  Energy as kcal/day and kcal/kg
Nutritional requirements and intake | From enrollment until 6 months after discharge
  Protein as gram/day and gram/kg
Nutritional requirements and intake | From enrollment until 6 months after discharge
  Fluids as ml/day and ml/kg
Nutritional requirements and intake | From enrollment until 6 months after discharge
  Total mineral an vitamin intake percentage of ADH
Feeding behaviour of the child | From enrollment until 6 months after discharge
  Questionnnaire CEBQ/BEBQ
Feeding behaviour of the child | From enrollment until 6 months after discharge
  Questionnnaire MCH-FS
Parental stress | From enrollment until 6 months after discharge
  Questionnaire LTO
Parental stress | From enrollment until 6 months after discharge
  Questionnaire PROMIS
Quality of Life of children and parents | From enrollment until 6 months after discharge
  Questionnaire CHU9D
Cost-effectiveness of tailored nutritional care | From enrollment until 6 months after discharge
  Questionnaire iMCQ
Cost-effectiveness of tailored nutritional care | From enrollment until 6 months after discharge
  Questionnaire iPCQ
Barriers and facilitators of implementation of the multidisciplinary support team | From enrollment until 6 months after discharge
  Interviews with parents

CONTACTS AND LOCATIONS:
Overall Officials: Sascha C Verbruggen, Principal Investigator — Erasmus Medical Center
Locations (1):
- ErasmusMC, Rotterdam, South Holland, Netherlands

IPD SHARING:
Plan to Share IPD: No